CLINICAL TRIAL: NCT02939391
Title: An Early Phase 2 Study of KW-6356 in Subject With Early Parkinson's Disease
Brief Title: A Study of KW-6356 in Subjects With Early Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6356-002
Record Dates: First submitted 2016-10-17; First posted 2016-10-20 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- KW-6356 Low Dose (Experimental): Oral administration
  Interventions: Drug: KW-6356
- KW-6356 High Dose (Experimental): Oral administration
  Interventions: Drug: KW-6356
- Placebo (Placebo Comparator): Oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KW-6356 — Oral administration
  Arms: KW-6356 Low Dose
Drug: KW-6356 — Oral administration
  Arms: KW-6356 High Dose
Drug: Placebo — Oral administration
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the effect of KW-6356 on motor symptoms in Parkinson's disease and the primary endpoint is the change from baseline in the MDS-UPDRS part III score between KW-6356 and placebo in subjects with early Parkinson's disease in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Subject fulfills the UK Parkinson's Disease Society brain bank clinical diagnostic criteria
* Parkinson's disease patients in Stages 1 to 3 on the Modified Hoehn and Yahr Scale
* MDS-UPDRS part III score of ≥ 15

Exclusion Criteria:

* Use of any CYP3A4/5-related drugs within 2 weeks prior to enrollment.
* Use of any of the specified antiparkinsonian drugs and dopamine antagonists during the specified period.
* Treatment with levodopa/DCI at any time in the past for a period of 4 weeks or more.
* Neurosurgical operation for Parkinson's disease (stereotactic surgery, deep brain stimulation or gamma knife), or treatment by transcranial magnetic stimulation (TMS).
* Either of the following criteria consecutively at screening and enrollment;

  * Resting Pulse > 100 bpm
  * Resting systolic blood pressure > 140 mmHg, or diastolic blood pressure > 90 mmHg
* Significant dementia or a Mini-Mental State Examination (MMSE) score of ≤ 23.
* Subject has a history or evidence of suicidal ideation (severity of 4 or 5) or any suicidal behavior based on an assessment with the Columbia-Suicide Severity Rating Scale (C-SSRS) at baseline.
* Anyone otherwise considered unsuitable for the study by the investigator or sub-investigator including those who are unable to communicate or to cooperate with the investigator or sub-investigator.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Movement disorder society-unified Parkinson's disease rating scale(MDS-UPDRS) partⅢ score | Up to 12 weeks after dosing

SECONDARY OUTCOMES:
Clinical global impression-improvement(CGI-I) score | Week 12
Patient global impression-improvement(PGI-I) score | Week 12
Change from baseline in the Parkinson's disease questionnaire-39(PDQ-39) total scores | Up to 12 weeks after dosing
Number and percentage of subjects with treatment-emergent adverse events | Up to 14 weeks after dosing
Profiles of pharmacokinetics of plasma KHK6356 concentration | 2, 4, 8 and 12 weeks after dosing
Change from baseline in the MDS-UPDRS subitem and total scores | Up to 12 weeks after dosing

CONTACTS AND LOCATIONS:
Locations (7):
- Japan (7):
  - Asahikawa, Hokkaido
  - Akashi, Hyōgo
  - Fujisawa, Kanagawa
  - Suita, Osaka
  - Nakano City, Tokyo
  - Setagaya City, Tokyo
  - Kyoto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maeda T, Kimura T, Sugiyama K, Yamada K, Hiraiwa R, Nishi M, Hattori N; 6356-002 study group. Randomized controlled trial of KW-6356 monotherapy in patients with early untreated Parkinson's disease. Parkinsonism Relat Disord. 2023 Dec;117:105907. doi: 10.1016/j.parkreldis.2023.105907. Epub 2023 Oct 31. PMID 37948832